CLINICAL TRIAL: NCT04396912
Title: Post-thyroidectomy Vocal Cord Paralysis Along With Hypocalcemia: Prospective, Matched-randomized Observational Cohort Compatible With STROBE Guidelines
Brief Title: Post-thyroidectomy Vocal Cord Paralysis Along With Hypocalcemia: STROBE - Guided Prospective Cohort
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ethem Unal, M.D., PhD, Associate Prof of Surgery & Surgic, MD, PhD, USMLE & IFSO-Certified, BCSS, Associated Professor of General Surgery and Surgical Oncology, Umraniye Education and Research Hospital
Other Study IDs: B.10.1TKH.4.34.H.GP0.01/1
Record Dates: First submitted 2020-05-15; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Iatrogenic Hypocalcemia; Iatrogenic Hypoparathyroidism; Vocal Cord Paralysis; Vocal Cord Paresis; Vocal Cord; Injury, Superficial; Thyroid Cancer, Papillary; Thyroid Cancer; Multinodular Goiter; Thyroid Neoplasms; Thyroid Nodule; Calcium Deficiency; PTH
Keywords: Total thyroidectomy
MeSH Terms: conditions — Vocal Cord Paralysis; Wounds and Injuries; Thyroid Cancer, Papillary; Thyroid Neoplasms; Thyroid Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control, s/p TT, without complication: Control (status/post-s/p total thyroidectomy-TT, without complication- demographics and BMI matched)
  Interventions: Procedure: Total thyroidectomy
- Experimental, s/p TT with only VCP: Experimental (s/p TT, with only vocal cord paralysis-VCP, uni or bilateral)
  Interventions: Procedure: Total thyroidectomy
- Experimental, s/p TT with only H: Experimental (s/p TT, with only hypocalcemia-H, transient or permanent)
  Interventions: Procedure: Total thyroidectomy
- Experimental, s/p TT with both VCP+H: Experimental (s/p TT, with both vocal cord paralysis-VCP and hypocalcemia-H);
  Subgroups:
  4.1. VCP (Permanent) + H (Permanent) 4.2. VCP (Transient) + H (Transient) 4.3. VCP (Permanent) + H (Transient) 4.4. VCP (Transient) + H (Permanent)
  Please answer:
  * Improvement in hypocalcemia also make a positive effect on voice? (any objective sign? Ca? PTH?)
  * Return of voice is parallel with the improvement in hypocalcemia? (any objective sign? Ca? PTH?
  Interventions: Procedure: Total thyroidectomy

INTERVENTIONS:
Procedure: Total thyroidectomy — Patients with thyroid diseases either benign (e.g. multinodular goitre) or malign (e.g. thyroid carcinoma) will be prepared for total thyroidectomy procedure and will be enrolled.

SUMMARY:
In the present study, the severity of recurrent laryngeal nerve injury (RLNI) and hypocalcemia (H) will be followed-up and the probable interrelation between them will be proposed considering the clinical situation of patients, e.g. improvement in hypocalcemia also make a positive effect on voice? (any objective sign? Ca? PTH?), return of voice is parallel with the improvement in hypocalcemia? Postoperative calcium (Ca), parathyroid hormone (PTH), regular vocal cord evaluations by ear-nose-throat (ENT) exams, deterioration-stability-improvement of clinical symptoms regarding both Ca metabolism and vocal cord function will be noted at regular intervals (postoperative day 1-3-first, weekly control/first month, monthly/first 6-month, 3-monthly/6-12 months) at outpatient controls. Serum Ca, PTH, ENT evaluation of vocal cords-noted.

DETAILED DESCRIPTION:
Total thyroidectomy is currently the preferred surgical treatment modality for both thyroid carcinomas and benign disorders such as multinodular goitre, since it minimizes the risk of recurrence and eliminates the complication risks of repeat or completion surgery. Vocal cord paralysis due to injury to recurrent laryngeal nerve (RLN) is the most dreaded complication of total thyroidectomy. The reported incidence of temporary RLN injury (RLNI) varies between 0 and 12 %, while the incidence of permanent RLNI has been reported to be much lower (0-3.5 %). In case of bilateral RLNI, respiratory distress and aspiration can develop rapidly and may result in mortality. Therefore, all precautions including close monitoring and tracheostomy should be undertaken without any delay. The best known technique to avoid injury to RLN is meticulous dissection of the nerve throughout its anatomic pathway. However, functional impairment of RLN is not visible macroscopically and intraoperative nerve monitoring (IONM) has been developed to monitor the nerve to avoid unnecessary dissection. Meticulous hemostasis can be achieved with harmonic sealing instrument, since improper hemostasis is known to increase the risk of RLNI. Despite the lack of evidence to support an advantage of IONM over the standard anatomic dissection of RLN, surgeons have adopted it in increasing ratios. The second most feared compliation of thyroidectomy is iatrogenic hypocalcemia. Transient symptomatic hypocalcemia after total thyroidectomy occurs in approximately 7% to 25% of cases, but permanent hypocalcemia is less common (0.4% to 13.8%). Size and invasion of tumor, operative trauma and vascular compromise determines the severity of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with total thyroidectomy indication, for either benign (e.g. multinodular goitre) or malign (e.g. thyroid carcinoma) thyroid disease
* >17 year-old
* Available for close follow-ups at outpatient clinic
* Available for close vocal cord exams

Exclusion Criteria:

* Patients with recurrent thyroid disease (benign/malign), prepared for a second operation
* Preferance of thyroid surgery other than total thyroidectomy

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with benign or malign thyroid diseases, eligable for total thyroidectomy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
s/p TT- normal (no complication) | June 01, 2020-June 01, 2021
  TT: total thyroidectomy
s/p TT+VCP | June 01, 2020-June 01, 2021
  VCP: vocal cord paralysis
s/p TT+H | June 01, 2020-June 01, 2021
  H: hypocalcemia
s/p TT+VCP+H | June 01, 2020-June 01, 2021
  Any improvement recorded? VCP? H? vice versa

SECONDARY OUTCOMES:
Improvement in vocal cord function /serum calcium | June 01, 2020-June 01, 2021
  VCP+H

CONTACTS AND LOCATIONS:
Overall Officials: Sema YUKSEKDAG, MD, Principal Investigator — Instructor in General Surgery; Ethem UNAL, MD, PhD, USMLE & IFSO-Certified, Board CSS, Study Chair — Assoc. Professor of General Surgery and Surgical Oncology
Locations (1):
- Umraniye Education and Research Hospital, Health Sciences University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study is open to high-volume INTERNATIONAL endocrine surgery centers, eager to join to present STROBE compatible observational study
  Available upon email requests@drethemunal@gmail.com
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From June 01, 2020, for 6 months
Access Criteria: Contact to drethemunal@gmail.com

REFERENCES:
- [Result] Cuschieri S. The STROBE guidelines. Saudi J Anaesth. 2019 Apr;13(Suppl 1):S31-S34. doi: 10.4103/sja.SJA_543_18. PMID 30930717
- [Result] Giulea C, Enciu O, Toma EA, Calu V, Miron A. The Tubercle of Zuckerkandl is Associated with Increased Rates of Transient Postoperative Hypocalcemia and Recurrent Laryngeal Nerve Palsy After Total Thyroidectomy. Chirurgia (Bucur). 2019 Sept-Oct;114(5):579-585. doi: 10.21614/chirurgia.114.5.579. PMID 31670633
- See also: STROBE guidelines — https://www.equator-network.org/reporting-guidelines/strobe/
- See also: Ethem Unal, MD, PhD (h-inde 18, i10-index 33) — https://scholar.google.com.tr/citations?user=6bFlCZwAAAAJ&hl=tr
- See also: VCP — https://www.journalagent.com/ejm/pdfs/EJM-33254-ORIGINAL_ARTICLE-YUKSEKDAG.pdf
- See also: TT complications — https://books.google.com.tr/books?id=MQX59bsB3CwC&pg=PA606&lpg=PA606&dq=recurrent+nerve+palsy+concurrent+hypocalcemia&source=bl&ots=H0OYiolBHv&sig=ACfU3U1_6EiiCEJ0mBCLikHDHHsoniUxkA&hl=tr&sa=X&ved=2ahUKEwiQpePr_rbpAhUlxMQBHYZdBWYQ6AEwAXoECAUQAQ#v=onepage&q=recurrent%20nerve%20palsy%20concurrent%20hypocalcemia&f=false